CLINICAL TRIAL: NCT02942082
Title: Clinical Evaluation for Post Bleaching Hypersensitivity Using Desensitizing Agent Before and /or After In-office Bleaching
Brief Title: Clinical Evaluation for Post Bleaching Hypersensitivity Using Desensitizing Agent During In-office Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Silvia Sabry, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBD-CU-2016-10-222
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Tooth Bleaching

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP oral care geldesensitizing agent (Experimental): a desensitizing agent will be applied on tooth before and /or after bleaching.
  Interventions: Other: ACP oral care gel
- glycrin (Placebo Comparator): glycrin will be applied on tooth before and /or after bleaching.
  Interventions: Other: glycrin

INTERVENTIONS:
Other: ACP oral care gel — a desensitizing agent will be applied on tooth before and/or after bleaching
  Arms: ACP oral care geldesensitizing agent
Other: glycrin — glycrin will be applied on tooth surface before and/or after bleaching
  Arms: glycrin

SUMMARY:
Evaluating the effect of a desensitizing agent on post-bleaching hypersensitivity.

DETAILED DESCRIPTION:
A randomized clinical trail will be done to evaluate the effect of a desensitizing agent ACP oral care gel in comparison to a control group on hypersensitivity after bleaching using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients must show no signs of spontaneous dental pain.
* Male or female patients between the ages of 18 to 40.
* Patients with good general and oral health.
* Patients having six caries-free maxillaryanterior teeth without restorations on the labial surfaces.
* Patients should have central incisors determined to be shade C2 or darker

Exclusion Criteria:

* Patient with spontaneous dental pain.
* Patient with anterior restorations or non carious cervical lesion.
* Patient having severe internal tooth discoloration (tetracycline stains, fluorosis, pulpless teeth), and bruxism habits.
* Tempro-mandibular joint problems involving symptomatic pain.
* Patients taking analgesics that could alter their normal pain perception level.
* Pregnant or breast feeding women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Post-bleaching hypersensitivity assessed using visual analogue scale | one month
  using visual analogue scale

SECONDARY OUTCOMES:
Tooth color assessed using value-ordered VITA® Classical Shade Guide | one month
  value-ordered VITA® Classical Shade Guide

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No